CLINICAL TRIAL: NCT05096754
Title: OCS Liver PROTECT Continued Access Protocol (CAP) Continuation Post-Approval Study
Status: Completed | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-LVR-02-PAS
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-05

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: OCS Liver — Transplant with an OCS preserved liver.

SUMMARY:
Post-approval observational study of subjects that were enrolled and transplanted in the OCS Liver PROTECT CAP.

ELIGIBILITY:
Inclusion Criteria:

* Subjects transplanted in the OCS Liver PROTECT CAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects transplanted in the OCS Liver PROTECT CAP
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Graft Survival | 24 Months
  Liver Graft Survival at 24 months post-transplant.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Scripps, La Jolla, California
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai, New York, New York
  - University of Texas Southwest, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia